CLINICAL TRIAL: NCT03298438
Title: Study About Annoucement of the Diagnosis of Neurofibromatosis 1 in de Novo Forms
Acronym: NF1
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: NF1
Record Dates: First submitted 2017-09-11; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Neurofibromatosis 1; Diagnoses Disease; Post Traumatic Stress Disorder
MeSH Terms: conditions — Neurofibromatosis 1; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurofibromatosis type 1 (NF1) is one of the most common autosomal dominant genetic disorders. The aim of our study was to evaluate post-traumatic stress disorder (PTSD) in patients and their families following the disclosure of sporadic NF1. Diagnosis of NF1 was retained according to NIH criteria, familial forms were excluded. The French version of the Impact of Event Scale-Revised was used for the diagnosis of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or more, or parent of a children
* Patient with a neurofibromatosis type 1 or parent of a children with a neurofibromatosis 1 in de novo form
* Followed for a neurofibromatosis type 1 de novo at the dedicated consultation in the University Hospital of Brest, since april 2013
* Agree to participate

Exclusion Criteria:

* Patients aged of 18 years old or lower
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients or parent of a children followed for a neurofibromatosis type 1 in de novo form
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Study post traumatic stress disorder secondary to annoucement of diagnosis of neurofibromatosis type 1 in de novo form | Day 1 after diagnosis of neurofibromatosis
  Questionnaire Impact of Event Scale

SECONDARY OUTCOMES:
Study methods of annoucement and feeling of patients with a questionnaire | Day 1 after diagnosis of neurofibromatosis
  Questionnaires about: methods of announcement (who? when? how?)
Genetical analyze | Day 1 after diagnosis of neurofibromatosis
  Genetical analyze
Psychological or psychiatrical impact | Day 1 after diagnosis of neurofibromatosis
  Psychological or psychiatrical impact
Information about NF1 | Day 1 after diagnosis of neurofibromatosis
  Questions about look for information about disease

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France